CLINICAL TRIAL: NCT03462992
Title: Peripheral Blood Monocytes as Predictive Marker for Colorectal Cancer Diagnosis: A Comparative Study of a Stool Based Versus Blood Based Screening Test
Acronym: MonoFIT+
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: DNAlytics (Industry)
Responsible Party: Principal Investigator, Hans Prenen, Professor, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: MonoFIT+
Record Dates: First submitted 2018-03-05; First posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FIT-positive individuals: Patients being positive to an FIT test performed in the context of the Flemish (Northern Belgium) colorectal cancer screening campaign. These patients are male and female between 56 and 74 years old.
  Interventions: Diagnostic Test: MonoMark

INTERVENTIONS:
Diagnostic Test: MonoMark — MonoMark (also known under the registered trademark ColonoKit), is a monocyte-based test using a transcriptomic signature and a mathematical predictive model aimed at discriminating between healthy individuals and CRC patients.

SUMMARY:
In this prospective study, the main goal is to evaluate the strength of Monomark -a monocyte-based transcriptomic test combined to a mathematical model- in patients with a positive FIT test. Therefore, in parallel to the routine FIT screening, blood samples will be harvested and the monocyte genetic profile will be determined. This fundamental study, will disclose the diagnostic power of a biomarker panel ("MonoMark") head to head with the well-established FIT diagnostic test, a core prerequisite for the routine use of this test as an alternative and more reliable CRC screening tool.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second leading cause of cancer death (approximately 9% of cancer deaths). In Belgium, a country with a population of 11,2 million people, every year 8600 patients get diagnosed with CRC. The cumulative risk is 5,1% for males and 3,5 % for females. Five-year survival of these patients is around 60%. Most colorectal cancers arise from polyps that progress from dysplasia to cancer. This adenoma - carcinoma sequence approximately takes several years. The slow transition from polyps to cancer allows opportunities to prevent CRC by removing polyps and early cancer. Although colonoscopic screening for CRC is currently the most reliable screening tool, the invasive nature and the incurred cost have hampered the wide application of this procedure. On the other hand, the fecal occult blood test (FOBT) and the most recently used fecal immunohistochemical test (FIT) are non-invasive screening tests that can be used prior to colonoscopy. However, they both lack the sensitivity or specificity required for an effective screening. Thus, there is a pressing need to identify specific non-invasive biomarkers for CRC early diagnosis.

Peripheral blood is an easily accessible tissue and therefore suitable for screening of disease biomarkers. Among the cells circulating in peripheral blood, monocytes are an interesting target as they represent a source of macrophages and dendritic cells, contributing to tumor growth, metastasis and angiogenesis as well as anti-tumor immune response.

Investigators from the Vlaams Instituut voor Biotechnologie (VIB) have over the years built an international network and team (UZ Leuven (Belgium), Jules Bordet Institute (Belgium), San Filippo Neri Hospital (Italy), University Hospital of Heidelberg (Germany)). With the initial aim to characterize different monocyte/macrophage phenotypes, the outstanding collaboration led to the development of an innovative test for the diagnosis of CRC that combines transcriptomic data with an efficient predictive model, the so-called "Monomark" test. In the Monomark study, VIB defined a genetic signature, which is induced specifically in circulating monocytes at early disease onset by soluble signals derived from transformed colon epithelium (in comparison to benign colon epithelium or other cancer histotypes). This gene signature was validated in a case-control study including 360 samples from the four European oncological centers with outstanding diagnostic accuracy, showing a sensitivity of about 90% and a specificity of about 95% (even when stratifying patients in stage I, II, III and IV) compared to other tests previously described or currently in use in the clinic (6,7). Moreover, preliminary data suggest the test can also detect relapse - an application that is being further developed.

Within this study investigators propose to further develop the Monomark test for the screening application, in order to maximize the interest from potential licensees. Investigators will need to show that the assay is superior to existing assays in casu the FOBT/FIT assays. Therefore, we will compare the sensitivity and specificity of this test head to head to the FIT stool test currently used in clinical screening for CRC. These findings will showcase Monomark's potential as a novel, non-invasive, cheap and safe assay for early detection of CRC, thus increasing the cure rate of CRC patients and reducing costs for the public health. The outstanding network built around the Monomark diagnostic platform will strongly support and speed up its validation and commercialization with specialized methodologies and analyses.

In this prospective study, the main goal is to evaluate the strength of the Monomark test in patients with a positive FIT test. Therefore, in parallel to the routine FIT screening, blood samples will be harvested and the monocyte genetic profile will be determined. This fundamental study, will disclose the diagnostic power of this biomarker panel head to head with the well-established FIT diagnostic test, a core prerequisite for the commercialization of the Monomark test as an alternative and more reliable CRC screening tool.

Currently, a Flemish screening project is ongoing in male and female patients between 56 and 74 years old. If patients have a positive stool test, they are advised to contact their general practitioner for planning of a colonoscopy. The goal is to avoid 400 deaths of colon cancer per year. In 2013, 248.970 patients were invited of which 49% send a stool sample to the lab. Of all the examined tests, 10.1% tested positive. However, only 5 to 10% of patients testing positive with the stool test are diagnosed with cancer. Therefore, the goal of this study is to discriminate with the monomark those patients with a high likelihood of having colon cancer.

At University Hospital Gasthuisberg (Leuven, Belgium) there are weekly about 5 patients with a positive stool test that are referred for a screening colonoscopy. It has been computed that 167 patients would be needed to evaluate the sensitivity and specificity of the Monomark test in patients with a positive stool test. To make sure that investigators can draw sound conclusions from this study, it is proposed to include 200 patients in total. In those patients it is planned to perform the blood based Monomark test. Therefore, during the first 12 months approximately 200 patients will be recruited whereas in the next 6 months all the molecular, bioinformatics and statistical analysis required will be performed to draw a robust and clear comparison.

The ultimate goal of this study is to provide solid data that the Monomark can be used as diagnostic tool and outperforms the current stool based diagnostic tests available on the market in order to screen more patients for early colon cancer and improve cure rate.

ELIGIBILITY:
Inclusion Criteria:

* Having participated to the Flemish (Northern Belgium) Colorectal Screening Campaign and, as a result, having a positive stool test (FIT) outcome.

Exclusion Criteria:

* None other than non-fulfillment of the inclusion criterion

Ages: 56 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Currently, a Flemish screening project is ongoing in male and female patients between 56 and 74 years old. If patients have a positive stool test, they are advised to contact their general practitioner for planning of a colonoscopy. The goal is to avoid 400 deaths of colon cancer per year. In 2013, 248.970 patients were invited of which 49% send a stool sample to the lab. Of all the examined tests, 10.1% tested positive. However, only 5 to 10% of patients testing positive with the stool test are diagnosed with cancer. Therefore, our goal is to discriminate with the monomark those patients with a high likelihood of having colon cancer. Patients of this study are patients who took part to this screening campaign and showed positive for the stool test.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2012-12-11 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2018-05-02 (Estimated)

PRIMARY OUTCOMES:
AUC of the MonoMark test | Within 1 year after recruitment completion.
  Area Under the ROC Curve (AUC) of the MonoMark test, comparing its predictions to the colonoscopy-confirmed status.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Prenen, MD, PhD, Principal Investigator — department of gastro-enterology, University Hospitals Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No